CLINICAL TRIAL: NCT07263750
Title: The Effect of Haptonomy Application for Primiparous Pregnant Women and Their Partners on Prenatal Attachment and Fear of Childbirth: A Randomized Controlled Study
Brief Title: Effect of Haptonomy on Prenatal Attachment and Fear of Childbirth in Primiparous Couples
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Sibel DİLMEN, Lecturer, Nigde Omer Halisdemir University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: OHU-DKH-SD-01
Record Dates: First submitted 2025-07-31; First posted 2025-12-04 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Fear of Childbirth; Prenatal Attachment
Keywords: fear of childbirth; pregnant; father; prenatal attachment; haptonomia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Haptonomy training will be provided to the experimental group within the childbirth class. Afterwards, the video-based haptonomy program will be sent via e-mail or WhatsApp. Couples will be asked to practice haptonomy exercises for five weeks, one 40-minute session per week.
  Interventions: Behavioral: Haptonomy
- control group (No Intervention): Standard of care Group The control group will not receive any treatment

INTERVENTIONS:
Behavioral: Haptonomy — Since there are no studies in the literature evaluating the effect of planned video modelling haptonomy on prenatal bonding and fear of childbirth in expectant mothers and fathers, it is believed that the results obtained from this study will contribute significantly to the literature by guiding and shedding light on future studies.
  Other Names: Haptonomy, as a field dealing with emotional contact through touch, describe the relationship between parents and the unborn baby.
  Arms: experimental group

SUMMARY:
This study was planned to evaluate the effect of haptonomy practice for primiparous pregnant women and their partners on prenatal attachment and fear of childbirth.

DETAILED DESCRIPTION:
Aim: This study was designed to evaluate the effect of haptonomy practice for primiparous pregnant women and their partners on prenatal attachment and fear of childbirth.

Methods: This randomized controlled experimental study will include primiparous pregnant women and their partners (36 couples in the experimental group and 36 couples in the control group) who apply to the childbirth education class of a public hospital in Turkey and are between 24-26 weeks of gestation.

The experimental group will receive haptonomy education in the childbirth class. Afterwards, a video-based haptonomy program will be delivered via e-mail or WhatsApp. Couples will be asked to perform haptonomy exercises once a week for 40 minutes over five weeks. No intervention will be applied to the control group.

Data will be collected before the intervention and at the end of the fifth week using the Personal Information Form, Prenatal Attachment Inventory (PAI), Wijma Delivery Expectancy/Experience Questionnaire Version A (W-DEQ A), Paternal-Fetal Attachment Scale (PFAS), and Fathers' Fear of Childbirth Scale (FFOC).

Data analysis will include frequency and percentage distributions, chi-square test, t-test, Mann-Whitney U test, repeated measures analysis, two-way ANOVA, Friedman test, and Cohen's d test.

ELIGIBILITY:
Inclusion Criteria:

* • At least a primary school graduate

  * Between the 24th and 26th weeks of pregnancy
  * According to calculations made by ultrasound based on the last menstrual period or, for pregnant women who do not know their last menstrual period, between the 24th and 26th weeks of pregnancy
  * Primiparous
  * No history of abortion/curettage
  * Planned/desired pregnancy
  * Desired baby gender
  * Living with spouse
  * Attended pregnancy classes
  * Able to use technology such as computers and mobile phones to watch videos
  * No barriers to understanding questions and responding
  * No previous training on fear of childbirth or prenatal bonding
  * Not having previously received education on haptonomy or practised haptonomy
  * Not undergoing infertility treatment
  * Being between the ages of 19 and 35

Exclusion Criteria:

* • Be at least 26 weeks pregnant

  * Live separately from spouse
  * Have an unplanned/unwanted pregnancy
  * Not want the baby to be of a specific gender
  * Not use technology
  * Be a high-risk pregnancy
  * Have previously received training on fear of childbirth and prenatal bonding
  * Having previously received training in haptonomy and practised haptonomy
  * Deciding to discontinue haptonomy practice after the study began and/or giving birth prematurely before completing the practice sessions

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2026-03-27 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Prenatal Attachment Inventory (PAI) | Baseline
  The PAI is a validated, explain thoughts, feelings, and situations experienced by woman during pregnancy and to determine the level of attachment to infant in prenatal period. Each item is of a four-point Likert type, with a score between 1 and 4. A minimum score of 21 and a maximum score of 84 can be obtained from the scale. Increase in the score obtained by pregnant indicates that level of attachment also increases.
Wijma Delivery Expectancy/Experience Questionnaire version A (W-DEQ-A) | Baseline
  The W-DEQ-A is a validated,to determine the level of birth fear experienced by pregnant women.Answers in the scale are numbered from 0 to 5 and are in a six-point Likert type. The minimum score that can be obtained from the scale is 0, and the maximum score is 165.
Paternal-Fetal Attachment Scale (PFAS) | Baseline
  PFAS is a validated scale used to determine the level of paternal-fetal attachment. The responses are rated on a four-point Likert scale ranging from 1 to 4. The minimum possible total score is 23, and the maximum is 92.
Fathers' Fear of Childbirth Scale (FFOC) | Baseline
  The FFOC is a validated instrument used to determine fathers' level of fear related to childbirth. The responses are rated on a five-point Likert scale ranging from 1 to 5. The minimum possible total score is 17, and the maximum is 85.

SECONDARY OUTCOMES:
Prenatal Attachment Inventory (PAI) | Week 5
  The PAI is a validated, explain thoughts, feelings, and situations experienced by woman during pregnancy and to determine the level of attachment to infant in prenatal period. Each item is of a four-point Likert type, with a score between 1 and 4. A minimum score of 21 and a maximum score of 84 can be obtained from the scale. Increase in the score obtained by pregnant indicates that level of attachment also increases.
Wijma Delivery Expectancy/Experience Questionnaire version A (W-DEQ-A) | Week 5
  The W-DEQ-A is a validated,to determine the level of birth fear experienced by pregnant women.Answers in the scale are numbered from 0 to 5 and are in a six-point Likert type. The minimum score that can be obtained from the scale is 0, and the maximum score is 165.
Paternal-Fetal Attachment Scale (PFAS) | Week 5
  PFAS is a validated scale used to determine the level of paternal-fetal attachment. The responses are rated on a four-point Likert scale ranging from 1 to 4. The minimum possible total score is 23, and the maximum is 92.
Fathers' Fear of Childbirth Scale (FFOC) | Week 5
  The FFOC is a validated instrument used to determine fathers' level of fear related to childbirth. The responses are rated on a five-point Likert scale ranging from 1 to 5. The minimum possible total score is 17, and the maximum is 85.

CONTACTS AND LOCATIONS:
Overall Officials: Nilüfer Tugut, Prof. Dr., Principal Investigator — Cumhuriyet University
Locations (1):
- Sivas Cumhuriyet University, Merkez, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ozbek H, Pinar SE. The effect of haptonomy applied to pregnant women on perceived stress, fear of childbirth, and prenatal attachment: randomized controlled experimental study. Curr Psychol. 2022 Jul 16:1-10. doi: 10.1007/s12144-022-03388-1. Online ahead of print. PMID 35874964